CLINICAL TRIAL: NCT05169112
Title: The Impact of Adjuvant Androgen Deprivation Following Radical Prostatectomy on Prostate Cancer Recurrence
Brief Title: Impact of Hormonal Therapy on Prostate Cancer Recurrence After Radical Prostatectomy
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: Tolmar Pharmaceuticals (Unknown)
Responsible Party: Principal Investigator, Rodney Breau, Dr., Ottawa Hospital Research Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Adjuvant ADT Pilot
Record Dates: First submitted 2021-03-01; First posted 2021-12-23 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Leuprolide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care (No Intervention): Standard of Care
- Standard of Care plus Androgen Deprivation Therapy (Lupron Depot) (Experimental): 22.5 mg intra-muscular injection of Lupron Depot every 3 months for 12 months (4 injections total)
  Interventions: Drug: Lupron Depot

INTERVENTIONS:
Drug: Lupron Depot — Patients randomized to receive androgen deprivation therapy (ADT) will receive 12 months of Lupron Depot (22.5 mg) administered every 3 months
  Arms: Standard of Care plus Androgen Deprivation Therapy (Lupron Depot)

SUMMARY:
Prostate cancer is the most common cancer in men and radical prostatectomy is the most frequent treatment for this disease. Unfortunately, approximately 40% of patients will develop recurrence after surgery, requiring additional salvage radiation. Salvage radiation after recurrence is successful in less than half of these men and most of those die from their disease. Measures to prevent recurrence are an important research priority for prostate cancer patients and their families. Hormonal therapy (androgen deprivation therapy; ADT) is routinely used to treat patients with metastases, but few clinical trials have examined if adjuvant ADT after surgery will prevent cancer recurrence. We aim to address this research oversight and test the hypothesis that for men at high risk of cancer recurrence, 1 year of ADT immediately after surgery will be safe and will significantly improve cancer outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. undetectable PSA (<0.02 ng/ml) within 16 weeks post-operative;
2. ≥25% predicted risk of PSA recurrence within 5 years of surgery (based on the Kattan nomogram)

Exclusion Criteria:

1. Unwilling to receive ADT;
2. previously received ADT;
3. lymph node metastases
4. allergy to any form of ADT

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2023-03-06 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2028-11 (Estimated)

PRIMARY OUTCOMES:
Rate of enrolment | 1 year
  Rate (patients/month) of enrolment

SECONDARY OUTCOMES:
Rate of enrolment per site | 1 year
  Rate (patients/month) of enrolment per site
Proportion of patients completing study intervention per-protocol | 1 year
  Proportion of patients completing study intervention per-protocol
Time to study start-up | 1 year
  Time to study start-up at each site
Completeness of study assessments | 1 year
  Proportion of study assessments completed per-protocol

CONTACTS AND LOCATIONS:
Locations (3):
- Canada (3):
  - Nova Scotia Health, Halifax, Nova Scotia
  - The Ottawa Hospital, Ottawa, Ontario
  - Centre universitaire de santé McGill - McGill University Health Centre, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No
N/A. IPD not planned to be shared